CLINICAL TRIAL: NCT04549480
Title: A PHASE 1, OPEN-LABEL, RANDOMIZED, 2-PERIOD, 2-SEQUENCE, CROSSOVER STUDY TO EVALUATE THE BIOEQUIVALENCE OF BOSUTINIB PEDIATRIC CAPSULE AND THE COMMERCIAL TABLET FORMULATIONS IN HEALTHY PARTICIPANTS UNDER FED CONDITION
Brief Title: Bioequivalence Study of Bosutinib Pediatric Capsule Relative to Commercial Tablet Under Fed Condition
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: B1871061; 2020-002782-34 (EudraCT Number)
Record Dates: First submitted 2020-09-08; First posted 2020-09-16 (Actual); Last update posted 2022-02-16 (Actual); Status verified 2022-02

CONDITIONS: Healthy Participants
Keywords: bosutinib,; bioequivalence,; Cmax,; AUC
MeSH Terms: interventions — bosutinib

STUDY DESIGN:
Masking Description: Open Label
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Bosutinib capsule (Experimental): Bosutinib pediatric capsule to healthy participants
  Interventions: Drug: Bosutinib capsule
- Bosutinib tablet (Active Comparator): Bosutinib tablet to healthy participants
  Interventions: Drug: Bosutinib tablet

INTERVENTIONS:
Drug: Bosutinib capsule — 100 mg dose of bosutinib pediatric capsule
  Arms: Bosutinib capsule
Drug: Bosutinib tablet — 100 mg dose of bosutinib tablet
  Arms: Bosutinib tablet

SUMMARY:
This study is intended to establish bioequivalence of the bosutinib age-appropriate capsule formulation to the commercial tablet formulation in healthy participants under fed condition. The comparison will be performed using the pharmacokinetic parameters that define the rate and extent of absorption, those are Cmax and AUC. A statistical analysis will be performed comparing these parameters calculated after administration of a single 100 mg dose with the tablet formulation (100 mg x 1) as the Reference treatment and the capsule formulation (100 mg x 1) as the Test treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Female participants of non childbearing potential and/or male participants must be 18 to 54 years of age, inclusive, at the time of signing the ICD.
2. Capable of giving signed informed consent as described in Appendix 1, which includes compliance with the requirements and restrictions listed in the ICD and in this protocol.

Exclusion Criteria:

1. Evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurological, dermatological, or allergic disease.
2. Any condition possibly affecting drug absorption.

Ages: 18 Years to 54 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 66 (Actual)
Dates: Start 2020-09-16 (Actual); Primary Completion 2021-01-15 (Actual); Study Completion 2021-01-15 (Actual)

PRIMARY OUTCOMES:
Area Under the Curve From Time Zero to Extrapolated Infinite Time [AUC (0-inf)] | 6 days
  Area Under the Curve From Time Zero to Extrapolated Infinite Time [AUC (0-inf)]
Maximum Observed Plasma Concentration (Cmax) | 6 days
  Maximum Observed Plasma Concentration (Cmax)

SECONDARY OUTCOMES:
Area Under the Curve From Time Zero to Last Quantifiable Concentration (AUClast) | 6 days
  Area Under the Curve From Time Zero to Last Quantifiable Concentration (AUClast)
Time to Cmax (Tmax) | 6 days
  Time to Cmax (Tmax)
Apparent Oral Clearance (CL/F) | 6 days
  Clearance of a drug is a measure of the rate at which a drug is metabolized or eliminated by normal biological processes.
Apparent Volume of Distribution (Vz/F) | 6 days
  Volume of distribution is defined as the theoretical volume in which the total amount of drug would need to be uniformly distributed to produce the desired plasma concentration of a drug.
Plasma elimination half-life (t1/2) | 6 days
  Plasma elimination half-life is the time measured for the plasma concentration to decrease by one half.

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (2):
- Netherlands (2):
  - PRA Health Sciences, Groningen
  - PRA Health Sciences Utrecht, Utrecht

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=B1871061